CLINICAL TRIAL: NCT06070337
Title: A Within-patient, Pilot Assessment of the Safety and Performance of H-Guard as a Priming Solution for Use in the Set-up of Blood Tubing Sets and Dialysers Prior to Use in Haemodialysis Patients
Brief Title: H-Guard Pilot Safety Evaluation in Haemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Invizius Limited (Industry)
Collaborators: Tailored Clinical Research Solutions (TCRS) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IH_001
Record Dates: First submitted 2023-03-29; First posted 2023-10-06 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2023-10

CONDITIONS: Renal Failure; Renal Insufficiency; Renal Disease
Keywords: Renal Failure; Haemodialysis; Renal; Kidney Failure; Dialysis
MeSH Terms: conditions — Renal Insufficiency; Kidney Diseases

STUDY DESIGN:
Intervention Model Description: This is a prospective, open label, pilot study of H-Guard® administered as a priming solution to both the blood tubing sets and dialyser of patients who are undergoing haemodialysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- H-Guard (Experimental): Participants receiving H-Guard Intervention.
  Interventions: Device: H-Guard

INTERVENTIONS:
Device: H-Guard — A novel Haemodialyser primer used for one treatment only

SUMMARY:
The purpose of this research study is to find out the safety and effectiveness of a new medical device called H-Guard.

During this research study, participants will receive the standard of care haemodialysis treatment, as decided by the treating doctor. Participants will be observed during 5-6 haemodialysis treatments throughout the course of the study. The only change to the treatment process, will be the use of the medical device (H-Guard) to prime the dialysis system, before one of the treatments.

Participants will have various blood tests taken throughout the course of the study for safety and research analysis.

DETAILED DESCRIPTION:
This prospective, open-label, study will be conducted in accordance with the requirements of EN ISO 14155, the Declaration of Helsinki (revised version of Edinburgh, Scotland 2000), Good Manufacturing Practice (GMP), Good Clinical Practice (GCP) and the current national regulations and guidelines, approved by both the local ethics committee and regulatory authority.

The study will be performed in a stable participant population who are on haemodialysis and who have a blood biomarker profile at screening, suggesting an increased risk of sensitivity to the haemodialysis dialyser and/or blood tubing sets (C3 deposition assay ratio ≤0.3 - measured immunologically using a C3 antibody in H-Guard vs human serum albumin coated ELISA plates). Participants will be recruited based on participation in a prior screening study and will attend a total of six-seven consecutive visits during the clinical trial

1. Screening [up to 30 days prior to the start of the clinical trial]
2. A non-interventional haemodialysis using standard priming solutions [Baseline - mid-week session: Day 0]
3. For WoCBP - a serum hCG test will be repeated between days 1-6 prior to intervention
4. A single haemodialysis using H-Guard to first prime the dialyser and tubing set [mid-week session: Day 7]
5. Followed by a further non-interventional haemodialysis without H-Guard [i.e. using standard priming solutions] [first haemodialysis post intervention]
6. A follow up visit 7 days post intervention to perform antibody analysis
7. Finally a follow up visit 14-21 days post intervention to perform antibody analysis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18 years and older at screening who have provided a signed and dated written informed consent
* Stable haemodialysis patients who are undergoing centre-based maintenance haemodialysis due to advanced kidney disease CKD stage 5, via arterio-venous fistula, graft or central venous catheter (i.e. with or without permanent vascular access)
* C3 deposition assay ratio ≤0.3 - measured immunologically using a C3 antibody in H-Guard vs human serum albumin coated ELISA plates
* Cytokine release assay - IL-6 concentrations following H-Guard vs Human Serum Albumin exposure must not exceed >50% and absence of significant Human Serum Albumin stimulated reactivity
* Willing and able to attend and comply with study visits and study related activities

Exclusion Criteria:

* Patients requiring haemodialysis for acute kidney injury on critical care (ITU)
* Patients unable or unwilling to comply with all trial procedures, e.g. blood sampling
* Patients with a likely survival prognosis of less than 6 months
* Patients who have been admitted for any acute hospital-based treatments in the last 6 weeks
* Patients on any medication which may interfere with the analysis of the biomarkers
* Current or history of use of anti-thrombotic therapy less than 7 days prior to screening.
* Currently active malignancy
* Currently receiving radiation, immunotherapy or chemotherapy
* Patients with active infection or receiving antibiotics within 30 days prior to screening
* Currently enrolled or has been enrolled in the last 30 days in another investigational device or drug study
* Known allergy or hypersensitivity to any component of the study device and/or medication to be used during the study.
* Patients lacking capacity to provide informed consent
* Pregnant or breastfeeding women
* Women of child-bearing potential (WoCBP)* who are unwilling to practice highly effective contraception** or undergo pregnancy tests at screening and during the study***
* Positive HIV and hepatitis B and C status, assessed from medical records only
* Patients with haematology or biochemistry results out of the normal reference range for this indication, assessed from medical records using test results obtained within 30 days of screening visit Any patients who are not deemed suitable for the study, as per the investigator's clinical opinion.

  * Pregnancy testing and contraception are not required for women not of child-bearing potential, including postmenopausal women or those with documented hysterectomy or bilateral oophorectomy. Postmenopausal women must be amenorrhoeic for at least 12 months in order not to be considered of childbearing potential. When postmenopausal status is uncertain, this will be confirmed by measurement of FSH.

    * Highly effective contraceptive measures include stable use of combined (oestrogen and progestogen containing) hormonal contraception (oral, intravaginal, transdermal) or progestogen-only hormonal contraception (oral, injectable, implantable) associated with inhibition of ovulation initiated 2 or more menstrual cycles prior to screening; intrauterine device (IUD); intrauterine hormone-releasing system (IUS); bilateral tubal ligation; vasectomized partner; and sexual abstinence***.

      * Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-10-19 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] when using H-Guard as a Priming Solution | Assessed from date of consent until the end of the study (day 28)
  Review of Adverse Events and Serious Adverse Event Frequency (All assessments)

SECONDARY OUTCOMES:
Assess the Presence of AOT Antibody Analysis 7 days Post Intervention | Assessed at visit 6 (day 14) [7 days after H-Guard intervention]
  Antibodies will be measured as ng/ml serum
Assess the Presence of AOT Antibody Analysis 14-21 days Post Intervention | Assessed at visit 7 (day 21-28) [14-21 days after H-Guard intervention]
  Antibodies will be measured as ng/ml serum
Changes in Biomarker Analysis (Coag) Prior to and Post Intervention (platelet count) | Assessed at visits screening, visit 4 (day 7) and visit 5 (day 10)
  Biomarkers of coagulation - Platelet count
Changes in Biomarker Analysis (Coag) Prior to and Post Intervention (wbc count) | Assessed at visits screening, visit 4 (day 7) and visit 5 (day 10)
  Biomarkers of coagulation - WBC count
Changes in Biomarker Analysis (Infl) Prior to and Post Intervention (CRP) | Assessed at visits screening, visit 4 (day 7) and visit 5 (day 10)
  Biomarkers of inflammation - CRP in mg/L
Changes in Biomarker Analysis (Infl) Prior to and Post Intervention (albumin) | Assessed at visits screening, visit 4 (day 7) and visit 5 (day 10)
  Biomarkers of inflammation - albumin in g/L
Analysis of Plasma AOT Proteins post intervention | Assessed at visit 4 (day 7) [H-Guard priming]
  Pharmacokinetic analysis of peak concentration in plasma (ng/ml plasma)
Measure of Dialysis Adequacy via Urea and Beta-2-Microglobulin Biomarkers | Assessed at visit 4 (day 7) [H-Guard priming] and visit 5 (day 10)
  To assess dialysis adequacy pre- and immediately post haemodialysis (H-Guard priming) (Urea and Beta 2 Microglobulin)

OTHER OUTCOMES:
To Analyse Participants Blood Biomarkers at Baseline Compared With Post H-Guard Intervention | Assessed at visits 2 (day 0), 4 (day 7) and 5 (day 10)
  Biomarkers for complement activation (Factor H), inflammation, coagulation and endothelial markers, WBC
Clinical Reported Endpoint Measure Analysis via Questionnaire | Immediately Post Haemodialysis with H-Guard used as a priming solution (day 7)
  Usability questionnaire completed by the treating user to confirm 'Ease of Use' Low to high.
Clinical Reported Endpoint Measure Analysis via Questionnaire | before, during and after H-Guard intervention (day 7) (visit 4)
  Usability questionnaire completed by the HCP user with the patient

CONTACTS AND LOCATIONS:
Overall Officials: Leonard Ebah, Principal Investigator — Manchester University NHS Foundation Trust; Magnus Nicolson, Study Director — Invizius Limited
Locations (1):
- Manchester Royal Infirmary, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
All data will be kept confidential and used only for the purpose of this study or future research about the device under investigation.